CLINICAL TRIAL: NCT06084169
Title: Single Center Post-Market Clinical Follow-Up (PMCF) Investigation for Assessing the Visual Performance of Hanita Lenses Intensity SL IOL in Comparison to Alcon Panoptix IOL
Brief Title: Investigation for Assessing the Visual Performance of Hanita Lenses Intensity SL IOL in Comparison to Alcon Panoptix IOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISL-01
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-10

CONDITIONS: Cataract
Keywords: IOL; Cataract; Hanita Lenses; Alcon; Intensity SL; Panoptix; Intra Ocular Lens
MeSH Terms: conditions — Cataract | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Intervention Model Description: The study will encompass a total of 58 patients:
  29 patients will be implanted bilaterally with Intensity SL IOL 29 patients will be implanted bilaterally with PanOptix IOL
Masking Description: Open Label Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensity SL IOL (Active Comparator): 29 patients will be implanted bilaterally with Intensity SL IOL
  Interventions: Device: Intra Ocular Lens (IOL) Implant
- Panoptix IOL (Active Comparator): 29 patients will be implanted bilaterally with PanOptix IOL
  Interventions: Device: Intra Ocular Lens (IOL) Implant

INTERVENTIONS:
Device: Intra Ocular Lens (IOL) Implant — Implantable intra ocular lens instead of the cataractous lens has been removed from the patient's eye
  Other Names: Panoptix Intra Ocular Lens (IOL) Implant

SUMMARY:
The goal of this clinical trial is to compare the visual performance between Intensity SL IOL and Panoptix IOL in men and women diagnosed with cataract who require cataract surgery procedure that meet the inclusion criteria and provide written informed consent will be enrolled in the study.

The main questions it aims to answer are:

1. To show non-inferiority in binocular distance corrected visual acuity for far, intermediate and near distances after Trifocal IOL implantation.
2. To show non-inferiority in the Defocus Curve measurement
3. To show non-inferiority in Contrast Sensitivity measurement
4. To show non-inferiority in patient satisfaction

Participants will attend a total of 10 study visits: 1 preoperative visit, 2 operations and 7 postoperative visits.

DETAILED DESCRIPTION:
This study is a single center, prospective, (1:1) randomized, unblinded, controlled study carried out in Germany according to Art. 74 MDR (PMCF study) or according to Art. 82 MDR / § 47 Para. 3 MPDG is carried out.

The lead investigator at the Heidelberg University Eye Clinic is Prof. Dr. Gerd U. Auffarth.

This study examines the visual performance of the trifocal Hanita Lenses Intensity SL IOL (study lens) compared to the trifocal Alcon PanOptix IOL (comparison lens) in bilaterally implanted patients. Clinical investigations including patient-reported results from the test group will be compared with those from the control group.

A total of approximately 58 patients will be included at 1 clinical center. Subjects participating in the study will attend a maximum of 10 study visits (1 preoperative, 2 operative and up to 7 postoperative) over a period of 3-7 months.

Only patients who have age-related cataracts will be included in the study. To participate in this study, patients must be at least 18 years old at the time of screening and a maximum preoperative corneal astigmatism of 1.0 D is permitted. All patients who would like to take part in this study will receive an information interview and further detailed study information in written form. Before a patient is admitted, he or she must sign a consent form.

The primary study endpoint is to investigate whether the binocular distance-corrected visual acuity achieved with the study lens for the distance, intermediate and near ranges is not statistically significantly inferior to the parameters achieved with the control lens.

The entire study including data processing will be carried out in accordance with EN ISO 14155:2020 Clinical Investigation of Medical Devices for Human Subjects, EN ISO 11979-7:2018: Clinical investigations of intraocular lenses for the correction of aphakia, EU MDR 2017/745, MEDDEV 2.7.1 rev. 4 Clinical Evaluation: A Guide for Manufacturers and Notified Bodies, MPDG:2020: Medical Device Law Implementation Act, as well as applicable local regulations and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Capability to understand and sign an IRB approved informed consent form and privacy authorization
* Age over 18 on the screening day
* Patients with bilateral age-related cataracts and planned bilateral cataract phacoemulsification combined Intraocular Lens implantation;
* Calculated IOL power is within range 15-30 Diopter (approximate range of axial lengths: 21-25.5mm)
* Normal corneas with corneal astigmatism below following value, measured by Biometer

  1. 1 D if with-the-rule (steep axis is vertical, between 60-120⁰)
  2. 0.4 D if against-the-rule (steep axis is horizontal, 0-30⁰ or 150-180⁰)
  3. 0.7 D if oblique (not one of the cases above)
* Post-operative best corrected distance visual acuity expected to be 0.3 logMAR or lower
* Patient motivated for trifocal IOL after screening by surgeon, willing and able to conform to the study requirements
* Fundus visualization is possible
* Absence of retinal or optic nerve diseases
* Clear intraocular media other than cataract
* When scheduling the first surgery, the patient shall commit to:

  1. Availability for the follow-up visits - 1 day, 1 week and 1 month after the first surgery
  2. Availability for the second surgery - one week to two months after the first surgery
  3. Availability for the follow-up visits - 1 day, 1 week, 1 month and 3 months after the second surgery

Exclusion Criteria:

* Difficulty for cooperation (distance from their home, general health conditions)
* Previous ocular/corneal surgery that may affect refraction accuracy or visual acuity.

  18 Protocol ID.: ISL-01 Version:2 Date: 20 Mar 2023
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* History or evidence of any ocular disease that may affect visual acuity (i.e. uncontrolled glaucoma, ocular injury, corneal pathologies, retinal pathologies in general and macular pathologies in particular, diabetic retinopathy, uveitis, aniridia or iris atrophy, vitreous pathologies (patients with vitreous separation or floaters can be included).
* Rubella cataract.
* Amblyopia
* Use of systemic or ocular medication that might affect vision
* Patients with, strabismus, former fruste keratoconus or keratoconus
* Usage of contact lenses during participation
* Any other ocular condition that may predispose a subject to future complications or contraindicate implantation of the trifocal lens.
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions)
* Pregnant, lactating, or planning to become pregnant during the course of the trial.
* Allergy or intolerance to required study medications (including antibiotic).
* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days.
* Traumatic cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Binocular distance corrected visual acuity | 3 months (90-120 days) post second eye operation
  To show non-inferiority in binocular distance corrected visual acuity for far, intermediate and near distances after Trifocal IOL implantation.
  Visual acuity will be performed by using ETDRS charts. All results will be expressed in logMAR. Visual acuity will be measured in photopic conditions.

SECONDARY OUTCOMES:
Defocus Curve | 3 months (90-120 days) post second eye operation
  To show non-inferiority in the Defocus Curve measurement by using ETDRS charts. The test will be performed using a phoropter to create defocus in 0.5D increments, starting from 1D to -4D relative to emmetropia so that the patient will be corrected for far vision.
Contrast Sensitivity | 3 months (90-120 days) post second eye operation
  To show non-inferiority in Contrast Sensitivity measurement by using VectorVision at mesopic and photopic conditions.
  Luminance for photopic conditions will be 85cd/m² and 5cd/m² for mesopic conditions. Small deviations are allowed. The working interval for photopic conditions is 75-95cd/m² and for mesopic conditions is 5-15cd/m².
Patient satisfaction | 3 months (90-120 days) post second eye operation
  To show non-inferiority in patient satisfaction by using the modified VF-14 questionnaire for quality of life, in addition to satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Auffarth Gerd U., Prof., Principal Investigator — Universitäts-Augenklinik Heidelberg International Vision Correction Research Centre (IVCRC)
Locations (1):
- Universitäts-Augenklinik Heidelberg International Vision Correction Research Centre (IVCRC), Heidelberg, Im Neuenheimer Feld, Germany

IPD SHARING:
Plan to Share IPD: No